CLINICAL TRIAL: NCT04938752
Title: An Open Label, Randomized, Single Dose, Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of DA 2811 in Healthy Subjects
Brief Title: Pharmacokinetics and Safety/Tolerability Profiles of DA-2811 in Healthy Subjects (DA-2811)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA2811_BE2_I
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence I (Experimental)
  Interventions: Drug: DA-2811; Drug: DA-2811-R
- Sequence II (Experimental)
  Interventions: Drug: DA-2811; Drug: DA-2811-R

INTERVENTIONS:
Drug: DA-2811 — single dose administration (one tablet once a day)
Drug: DA-2811-R — single dose administration (one tablet once a day)

SUMMARY:
This is the phase I study to evaluate the pharmacokinetics and safety of DA-2811 and DA-2811-R after a single oral dose in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* BMI between 18.5 and 29.9 kg/m2 and weigh at least 50 kg
* Volunteer who totally understands the progress of this clinical trial, make decision by his or her free will, and signed a consent form to follow the progress

Exclusion Criteria:

* Volunteer who has present or past history of clinically significant cardiovascular, respiratory, urinary, gastrointestinal, hepatic, renal, skin, immunological, musculoskeletal, endocrinal, neurological, psychiatric and/or hematological disease

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
AUClast | pre-dose~48 hours post-dose
  Area under the plasma concentration-time curve from time zero to time the last quantifiable time
Cmax | pre-dose~48 hours post-dose
  Maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Chung JaeYong, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam-si, South Korea